CLINICAL TRIAL: NCT01572298
Title: A Prospective Study: Alveolar Ridge Augmentation Using Tenting Screws, Acellular Dermal Matrix and Combination Particulate Grafts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20120108H
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2015-10

CONDITIONS: Dental Alveolus; Oral Surgical Procedures, Preprosthetic
MeSH Terms: interventions — Transplantation, Homologous; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allograft alone (Active Comparator): guided bone regeneration with allograft alone (includes tenting screws and overlying allograft membrane material)
  Interventions: Device: allograft alone
- allograft with autograft (Experimental): guided bone regeneration with allograft and autograft combined (includes tenting screws and overlying allograft membrane material)
  Interventions: Device: allograft with autograft

INTERVENTIONS:
Device: allograft alone — use of MinerOss allograft plus Alloderm GBR membrane and tenting screws
  Arms: allograft alone
Device: allograft with autograft — use of a combined autogenous graft and MinerOss allograft plus Alloderm GBR membrane and tenting screws
  Arms: allograft with autograft

SUMMARY:
When a tooth or teeth are extracted, a defect in the bony ridge often forms. This loss of bone may make it impossible to place a dental implant. Guided bone regeneration procedures are used to re-establish a bone dimension sufficient to place a dental implant. The primary objective of the study is to determine whether there is any difference in the gain of horizontal alveolar ridge width following guided bone regeneration surgery using a combined autogenous/allogenic particulate bone graft versus a particulate allograft alone. Autogenous bone has historically been considered the gold standard for alveolar ridge grafting; however, other materials including allografts and xenografts have also been used with excellent results. This study evaluates the potential benefits, or lack thereof, for using a combined autogenous/allograft approach versus an allograft alone. The investigators will clinically evaluate the efficacy of this technique and determine the difference in bone formation between groups following healing at 5 months by observing bone growth relative to heads of the tenting screws placed horizontally in the locations of greatest defect in the alveolar ridge. A biopsy of the healed site will be taken at the time of implant placement. The null hypothesis is that there will be no difference in the amount of horizontal ridge width gain at 5 months post-grafting between the two different grafting materials (allograft alone versus allograft combined with autogenous bone). Furthermore, the null hypothesis is that histologically, the combination graft (MinerOss®/particulate autograft) will have a similar percentage of vital bone present at 5 months compared to the allograft-alone group (MinerOss®).

DETAILED DESCRIPTION:
Guided bone regeneration procedures are used to re-establish a bone dimension sufficient to place a dental implant. The primary objective of the study is to determine whether there is any difference in the gain of horizontal alveolar ridge width following guided bone regeneration surgery using a combined autogenous/allogenic particulate bone graft versus a particulate allograft alone. Autogenous bone has historically been considered the gold standard for alveolar ridge grafting; however, other materials including allografts and xenografts have also been used with excellent results. This study evaluates the potential benefits, or lack thereof, for using a combined autogenous/allograft approach versus an allograft alone. The investigators will clinically evaluate the efficacy of this technique and determine the difference in bone formation between groups following healing at 5 months by observing bone growth relative to heads of the tenting screws placed horizontally in the locations of greatest defect in the alveolar ridge. A biopsy of the healed site will be taken at the time of implant placement. The null hypothesis is that there will be no difference in the amount of horizontal ridge width gain at 5 months post-grafting between the two different grafting materials (allograft alone versus allograft combined with autogenous bone). Furthermore, the null hypothesis is that histologically, the combination graft (MinerOss®/particulate autograft) will have a similar percentage of vital bone present at 5 months compared to the allograft-alone group (MinerOss®).

ELIGIBILITY:
Inclusion Criteria:

* subject with a partially edentulous ridge of the maxilla or mandible with at least one tooth-span in length and inadequate buccolingual dimension for dental implant placement as measured clinically and radiographically
* live within "catchment area" of 50 mile radius from San Antonio

Exclusion Criteria:

* unstable systemic disease (such as compromised immune system)
* patient taking steroids or other medications affecting bone metabolism
* patient with history of radiation therapy to head & neck
* history of previous ridge augmentation procedure or pathology at local jaw site
* smokers who smoke > 10 cigarettes per day

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Mealey, DDS, MS, Principal Investigator — Univ of Texas Health Science Center at San Antonio
Locations (1):
- University of texas Health Science Center Dental School at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Allograft Alone: guided bone regeneration with allograft alone (includes tenting screws and overlying allograft membrane material)
  allograft alone (MinerOss allograft plus Alloderm GBR membrane): use of MinerOss allograft plus Alloderm GBR membrane and tenting screws
- Allograft Combined With Autograft: guided bone regeneration with allograft and autograft combined (includes tenting screws and overlying allograft membrane material)
  allograft combined wtih autograft (combined autogenous graft and MinerOss allograft plus Alloderm GBR membrane): use of a combined autogenous graft and MinerOss allograft plus Alloderm GBR membrane and tenting screws
Period: Overall Study
Arm/Group | Allograft Alone | Allograft Combined With Autograft
Started | 14 | 13
Completed | 12 | 12
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allograft Alone | Allograft Combined With Autograft | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.8) | 47.5 (14.5) | 48.9 (12.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Gain in Horizontal Ridge Dimension
Time Frame: 5 months after surgery
Measure: Mean (Standard Deviation); unit: gain in ridge width (mm)
Arm/Group | Allograft Alone | Allograft Combined With Autograft
Number analyzed (Participants) | 12 | 11
gain in ridge width (mm) | 3.33 (0.83) | 3.09 (0.63)

2. Secondary Outcome: Percentage of New Bone Formation (Histologic)
Time Frame: 5 months after surgery
Population: No data were collected for this outcome
Arm/Group | Allograft Alone | Allograft With Autograft
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Allograft Alone | Allograft Combined With Autograft
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes